CLINICAL TRIAL: NCT05138796
Title: A Phase 1, Randomized, Double-Blind, Single- and Multiple-Ascending-Dose Study Evaluating the Safety, Tolerability, Food-Effect and Pharmacokinetics of TP-05 in Healthy Subjects
Brief Title: A Pharmacokinetic Study of TP-05 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tarsus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Basic Science
Other Study IDs: TRS-013
Record Dates: First submitted 2021-07-22; First posted 2021-12-01 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Healthy
MeSH Terms: interventions — lotilaner

STUDY DESIGN:
Intervention Model Description: Part 1: a randomized, double-blind, single ascending dose (SAD) with Cohort 1-4 administered on a full stomach and Cohort 5 administered after a period of fasting Part 2: a randomized, double-blind, multiple ascending dose (MAD) escalation with Cohort 6-8 administered on a full stomach.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The investigators, study coordinators, study subjects, and the sponsor will be blinded to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- TP-05 SAD (Experimental): Single dose of TP-05 (lotilaner oral capsules) at 4 dose levels in ascending order
  Interventions: Drug: TP-05 (lotilaner oral capsules)
- Placebo SAD (Experimental): Single dose of Placebo
  Interventions: Drug: Placebo
- TP-05 MAD (Experimental): Four doses of TP-05 (lotilaner oral capsules) at 3 dose levels in ascending order
  Interventions: Drug: TP-05 (lotilaner oral capsules)
- Placebo MAD (Experimental): Four doses of Placebo
  Interventions: Drug: Placebo
- TP-05 Fasted (Experimental): Single dose of TP-05 (lotilaner oral capsules) in a fasted state
  Interventions: Drug: TP-05 (lotilaner oral capsules)
- Placebo Fasted (Experimental): Single dose of placebo in a fasted state
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TP-05 (lotilaner oral capsules) — TP-05 (lotilaner oral capsules)
  Arms: TP-05 Fasted; TP-05 MAD; TP-05 SAD
Drug: Placebo — Placebo to match TP-05 (lotilaner oral capsules)
  Arms: Placebo Fasted; Placebo MAD; Placebo SAD

SUMMARY:
A Phase 1, Randomized, Double-Blind, Single- and Multiple-Ascending Dose Study Evaluating the Safety, Tolerability, Food-Effect and Pharmacokinetics of TP-05 in Healthy Subjects

DETAILED DESCRIPTION:
This Phase 1 study is a randomized, double-blind, single- and multiple-ascending dose trial to evaluate the safety, tolerability, food-effect, and pharmacokinetics of TP-05 in healthy subjects. Subjects will be enrolled in 5 sequential, ascending single dose cohorts and 3 multiple, ascending dose cohorts. Dose escalation will be approved by a safety monitoring committee before beginning the next cohort. The Safety Review Committee (SRC) will evaluate if any dose-limiting adverse events (AEs) through Day 15 (in Cohorts 1-5) or through Day 36 (in Cohorts 6-8) occurred in a cohort before proceeding to dosing in the next dose level. In addition, the SRC will review selected PK parameters after selected cohorts. Skin punch biopsies, and venous, capillary, and urine samples may be collected at various timepoints for pharmacokinetic analysis. Safety assessments include monitoring of adverse events, clinical laboratory testing, vital sign measurements, physical examinations, and ECGs. A blood sample may also be collected to evaluate tick mortality upon exposure.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form (ICF)
2. Have no clinically significant diseases captured in the medical history or evidence of clinically significant findings on the physical examination (including vital signs) and/or ECG, as determined by an investigator

Exclusion Criteria:

1. Female who is pregnant or lactating
2. Presence or history of significant gastrointestinal, metabolic, liver or kidney disease, or surgery that may affect drug bioavailability (excluding appendectomy and cholecystectomy)
3. History of significant cardiovascular, pulmonary, hematologic, neurological, psychiatric, endocrine, immunologic, or dermatologic disease
4. Have a history of a malignancy (or active malignancy), with the exception of treated basal cell or squamous cell carcinoma
5. Use of any prescription drugs (with the exception of hormonal contraceptives or hormone replacement therapy) within 14 days prior to or use of any over-the-counter drugs in the 7 days prior to the first study drug administration
6. Positive urine alcohol test result and/or drugs of abuse at Screening or prior to the first drug administration (including cotinine, cannabinoids, amphetamines, barbiturates, cocaine, opiates, phencyclidine and benzodiazepines)
7. Positive test results for HIV-1/HIV-2 Antibodies, Hepatitis B surface Antigen (HBsAg) or Hepatitis C Antibody (HCVAb)
8. Treatment with an investigational drug within 30 days or 5 times the half-life (whichever is longer) prior to Screening
9. Blood donation (excluding plasma donation) of approximately 500 mL within 56 days prior to Screening
10. Plasma donation within 7 days prior to screening

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-07-25 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events (TEAEs) | up to 151 days
  Evaluate the safety of TP-05 through the incidence rate of TEAEs
Clinically significant changes from Baseline chemistry laboratory tests | up to 151 days
  Evaluate the safety of TP-05 through clinically significant changes from Baseline chemistry laboratory tests
Clinically significant changes from Baseline hematology laboratory tests | up to 151 days
  Evaluate the safety of TP-05 through clinically significant changes from Baseline hematology laboratory tests
Clinically significant changes from Baseline general appearance | up to 151 days
  Evaluate the safety of TP-05 through clinically significant changes from Baseline general appearance
Clinically significant changes from Baseline physical examination of head, ears, nose, and throat | up to 151 days
  Evaluate the safety of TP-05 through clinically significant changes from Baseline physical examinations of head, ears, nose, and throat
Clinically significant changes from Baseline physical examination of neck (thyroid) | up to 151 days
  Evaluate the safety of TP-05 through clinically significant changes from Baseline physical examinations of neck (thyroid)
Clinically significant changes from Baseline physical examination of respiratory system | up to 151 days
  Evaluate the safety of TP-05 through clinically significant changes from Baseline physical examinations of respiratory system
Clinically significant changes from Baseline physical examination of cardiovascular system | up to 151 days
  Evaluate the safety of TP-05 through clinically significant changes from Baseline physical examinations of cardiovascular system
Clinically significant changes from Baseline physical examination of gastrointestinal system | up to 151 days
  Evaluate the safety of TP-05 through clinically significant changes from Baseline physical examinations of gastrointestinal system
Clinically significant changes from Baseline physical examination of neurological system | up to 151 days
  Evaluate the safety of TP-05 through clinically significant changes from Baseline physical examinations of neurological system
Clinically significant changes from Baseline physical examination of musculoskeletal system (extremities) | up to 151 days
  Evaluate the safety of TP-05 through clinically significant changes from Baseline physical examination of musculoskeletal system (extremities)
Clinically significant changes from Baseline physical examination of skin | up to 151 days
  Evaluate the safety of TP-05 through clinically significant changes from Baseline physical examination of skin
Clinically significant changes from Baseline vital signs | up to 151 days
  Evaluate the safety of TP-05 through clinically significant changes from Baseline vital signs (including temperature [degrees Celsius], pulse rate [beats per minute], respiration rate [breaths per minute], and changes in systolic and diastolic blood pressure [mmHg])
Clinically significant changes from Baseline vital signs (temperature [degrees Celsius]) | up to 151 days
  Evaluate the safety of TP-05 through clinically significant changes from Baseline vital signs including temperature [degrees Celsius]
Clinically significant changes from Baseline vital signs (pulse rate [beats per minute]) | up to 151 days
  Evaluate the safety of TP-05 through clinically significant changes from Baseline vital signs including pulse rate [beats per minute]
Clinically significant changes from Baseline vital signs (respiration rate [breaths per minute]) | up to 151 days
  Evaluate the safety of TP-05 through clinically significant changes from Baseline vital signs including respiration rate [breaths per minute]
Clinically significant changes from Baseline vital signs (systolic and diastolic blood pressure [mmHg]) | up to 151 days
  Evaluate the safety of TP-05 through clinically significant changes from Baseline vital signs including changes in systolic and diastolic blood pressure [mmHg])
Clinically significant changes from Baseline electrocardiograms (ECGs) | up to 151 days
  Evaluate the safety of TP-05 through clinically significant changes from Baseline ECGs (including changes in mean ventricular rate [beats/min], pulse rate [msec], QRS duration [msec], QT interval [msec], QTcF interval [msec])

SECONDARY OUTCOMES:
Exposure and PK of lotilaner in whole blood | up to 151 days
  PK parameters for whole blood sampling methods following dose administration will be evaluated and include Cmax at various times
Exposure and PK of lotilaner in whole blood | up to 151 days
  PK parameters for whole blood sampling methods following dose administration will be evaluated and include Tmax at various times
Exposure and PK of lotilaner in whole blood | up to 151 days
  PK parameters for whole blood sampling methods following dose administration will be evaluated and include Tlag at various times
Exposure and PK of lotilaner in whole blood | up to 151 days
  PK parameters for whole blood sampling methods following dose administration will be evaluated and include AUC0-168 at various times
Exposure and PK of lotilaner in whole blood | up to 151 days
  PK parameters for whole blood sampling methods following dose administration will be evaluated and include AUC0-2880 at various times
Exposure and PK of lotilaner in whole blood | up to 151 days
  PK parameters for whole blood sampling methods following dose administration will be evaluated and include AUC0-t at various times
Exposure and PK of lotilaner in whole blood | up to 151 days
  PK parameters for whole blood sampling methods following dose administration will be evaluated and include AUC0-inf at various times
Exposure and PK of lotilaner in whole blood | up to 151 days
  PK parameters for whole blood sampling methods following dose administration will be evaluated and include CL/F at various times
Exposure and PK of lotilaner in whole blood | up to 151 days
  PK parameters for whole blood sampling methods following dose administration will be evaluated and include Vz/F at various times
Exposure and PK of lotilaner in whole blood | up to 151 days
  PK parameters for whole blood sampling methods following dose administration will be evaluated and include eff at various times
Exposure and PK of lotilaner in whole blood | up to 151 days
  PK parameters for whole blood sampling methods following dose administration will be evaluated and include Thalf at various times
Exposure and PK of lotilaner in whole blood | up to 151 days
  PK parameters for whole blood sampling methods following dose administration will be evaluated and include λz at various times
Exposure and PK of lotilaner in whole blood | up to 151 days
  PK parameters for whole blood sampling methods following dose administration will be evaluated and include AUC%extrap at various times
Exposure and PK of lotilaner in whole blood | up to 151 days
  PK parameters for whole blood sampling methods following dose administration will be evaluated and include MRT0-t at various times
Exposure and PK of lotilaner in whole blood | up to 151 days
  PK parameters for whole blood sampling methods following dose administration will be evaluated and include Rac at various times
Exposure and PK of lotilaner in whole blood | up to 151 days
  PK parameters for whole blood sampling methods following dose administration will be evaluated and include Ctrough at various times
Urine exposure and renal PK of lotilaner | 3 days
  PK parameters for urine sampling methods will be evaluated and include Ae.
Urine exposure and renal PK of lotilaner | 3 days
  PK parameters for urine sampling methods will be evaluated and include fe.
Urine exposure and renal PK of lotilaner | 3 days
  PK parameters for urine sampling methods will be evaluated and include CLr0-48.
Impact of fasting on the PK of lotilaner | up to 151 days
  PK parameters will be evaluated for lotilaner following dosing with food and under fasting conditions. Parameters include Cmax at various times
Impact of fasting on the PK of lotilaner | up to 151 days
  PK parameters will be evaluated for lotilaner following dosing with food and under fasting conditions. Parameters include Tmax at various times
Impact of fasting on the PK of lotilaner | up to 151 days
  PK parameters will be evaluated for lotilaner following dosing with food and under fasting conditions. Parameters include Tlag at various times
Impact of fasting on the PK of lotilaner | up to 151 days
  PK parameters will be evaluated for lotilaner following dosing with food and under fasting conditions. Parameters include AUC0-168 at various times
Impact of fasting on the PK of lotilaner | up to 151 days
  PK parameters will be evaluated for lotilaner following dosing with food and under fasting conditions. Parameters include AUC0-2880 at various times
Impact of fasting on the PK of lotilaner | up to 151 days
  PK parameters will be evaluated for lotilaner following dosing with food and under fasting conditions. Parameters include AUC0-t at various times
Impact of fasting on the PK of lotilaner | up to 151 days
  PK parameters will be evaluated for lotilaner following dosing with food and under fasting conditions. Parameters include AUC0-inf at various times
Impact of fasting on the PK of lotilaner | up to 151 days
  PK parameters will be evaluated for lotilaner following dosing with food and under fasting conditions. Parameters include CL/F at various times
Impact of fasting on the PK of lotilaner | up to 151 days
  PK parameters will be evaluated for lotilaner following dosing with food and under fasting conditions. Parameters include Vz/F at various times
Impact of fasting on the PK of lotilaner | up to 151 days
  PK parameters will be evaluated for lotilaner following dosing with food and under fasting conditions. Parameters include Thalf at various times
Impact of fasting on the PK of lotilaner | up to 151 days
  PK parameters will be evaluated for lotilaner following dosing with food and under fasting conditions. Parameters include λz at various times
Impact of fasting on the PK of lotilaner | up to 151 days
  PK parameters will be evaluated for lotilaner following dosing with food and under fasting conditions. Parameters include AUC%extrap at various times
Impact of fasting on the PK of lotilaner | up to 151 days
  PK parameters will be evaluated for lotilaner following dosing with food and under fasting conditions. Parameters include MRT0-t at various times
Impact of fasting on the PK of lotilaner | up to 151 days
  PK parameters will be evaluated for lotilaner following dosing with food and under fasting conditions. Parameters include Rac at various times
Impact of fasting on the PK of lotilaner | up to 151 days
  PK parameters will be evaluated for lotilaner following dosing with food and under fasting conditions. Parameters include Ctrough at various times

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Lim, Study Director — Tarsus Pharmaceuticals
Locations (1):
- Altasciences, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No